CLINICAL TRIAL: NCT04405050
Title: Randomized Clinical Trial to Compare Restrata and Negative Pressure Wound Therapy (NPWT) to Heal Complex Diabetic Foot Wounds
Brief Title: RCT to Compare Restrata and NPWT to Heal Complex DFUs
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Project Never Initiated - no human subjects were enrolled and no data regarding humans was collected or studied.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Acera Surgical, Inc. (Industry)
Responsible Party: Principal Investigator, Larry Lavery, Professor and Director of Research, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0268
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Wound
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: This study is a prospective, 2-arm parallel assignment, randomized clinical trial to compare Restrata and NPWT in patients with complex diabetic foot ulcers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Restrata (Active Comparator): Treated with Restrata
  Interventions: Device: Restrata
- NPWT (Active Comparator): Treated with NPWT (Negative Pressure Wound Therapy)
  Interventions: Device: Negative Pressure Wound Therapy (NPWT)

INTERVENTIONS:
Device: Restrata — Restrata® is a novel synthetic nanofabricated scaffold (Restrata Wound Matrix (RWM), Acera Surgical, St. Louis, Missouri) has been developed which is a sterile, single-use device intended for use in the local management of wounds. The RWM is a soft, white, conformable, non-friable, absorbable matrix that acts as a protective covering for wound defects, providing a moist environment for the body's natural healing process to occur (Figure 2). The RWM is made from synthetic biocompatible materials and was designed to include a fibrous structure with high porosity, similar to native ECM. As a viable wrap for surgical procedures, Restrata conforms to injured tissue, can be sutured, and is arthroscopic and robotic procedure friendly.
  Arms: Restrata
Device: Negative Pressure Wound Therapy (NPWT) — Negative Pressure Wound Therapy (NPWT) has dramatically changed the care of complex foot wounds. Compared to standard wound care, patients with diabetic foot wounds that are treated with NPWT are 5.9 times more likely to heal and 4.4 times less likely to require amputation. NPWT involves the delivery of sub-atmospheric pressure through a vacuum pump connected to a specialized dressing to maintain a closed environment. NPWT increases perfusion to the wound, accelerates granulation tissue formation, reduces edema, and reduces bio-burden
  Arms: NPWT

SUMMARY:
The purpose of this study is to compare the efficacy of Restrata compared to Negative Pressure Wound Therapy (NPWT) to heal complex diabetic foot wounds.

DETAILED DESCRIPTION:
Screening

1. Explain purpose and nature of the study and obtain signature on the informed consent document.
2. Screen the subject against protocol inclusion and exclusion criteria, including all pertinent tests, including pregnancy test if needed.

Baseline (may be done as same day as screening procedures)

1. Obtain general medical history and demographic information and social history
2. Complete a physical examination, body weight, height, and vital signs, including measurement of resting heart rate, respiratory rate, and blood pressure while seated.
3. Select target study ulcer
4. Obtain complete history pertinent to DFU disease including duration of the target ulcer, previous and current treatment.
5. Perform debridement and obtain tissue collection (3 tissue and 1 bone if applicable).
6. Perform standardized photography and measurement of the study wound (eKare or available camera with ruler). Assess the post-debridement ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device (eKare, Fairfax, VA).
7. Perform hyperspectral imaging of dorsal and plantar aspects of the foot.
8. Perform neuropathy assessment (monofilament, VPT)
9. Skin perfusion pressure (Sensilase)
10. Collect all relevant concomitant medication (antibiotics, steroids, and diabetes medications)
11. Complete questionnaires
12. Place Restrata and dress wound or apply NPWT therapy.
13. Submit subject stipend

Therapy/Treatment Phase

Study Visit 1-11:

1. Assess target ulcer (if wound has closed, document as such, skip to END OF STUDY VISIT (EOS).
2. Document time on/off NPWT if applicable.
3. If Restrata is removed, assess the ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device - if the wound is deemed healed by the physician, skip to EOS visit.
4. Perform hyperspectral imaging of the dorsal and plantar aspects of the foot if wound is active or healed.
5. Debride wound if indicated. Re-measure wound if surgical debridement is performed prior to dressing the wound
6. Collect all relevant concomitant medication.
7. If wound is not healed, redress the wound with Restrata dressing (if removed for debridement) or NPWT.
8. Disburse subject stipend
9. Note: at week 3, if wound is not ready for surgical closure, remove Restrata and replace with new piece of Restrata (per randomization schedule)
10. Assess for AE/SAEs and/or follow up on previous AE/SAEs.

Study Visit Closed

1. When a study wound has closed, we will perform the EOS evaluation.
2. If a wound has closed, the patient will enter the follow-up phase of the study.

Study Visit 12/EOS:

1. If the study wound closes prior to the 12-week study mark, subjects will perform EOS visit at the time of wound closure.
2. Assess target ulcer.
3. If wound has not closed, assess the ulcer area (cm2), perimeter (cm), and greatest depth (cm) using the inSight device.
4. Perform hyperspectral imaging of the dorsal and plantar aspects of the foot if wound is active or healed.
5. If wound has not closed, redress the wound per physician-directed standard of care.
6. Perform EOS visit documentation
7. Complete questionnaires
8. Follow up on AE/SAEs that have not yet been resolved.

Study Visit Follow-up

1. If the wound heals during the treatment phase or if the wound is not healed after 12 weeks, data from their electronic medical record will be evaluated to identify healing, time to heal, adverse events related to the wound.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a diabetes mellitus
* Men/women ≥21 years old
* Post-operative foot or ankle wounds sized < 15cm
* ABI ≥0.5 or toe pressures >30 mmHg
* Wounds indicated for treatment with NPWT

Exclusion Criteria:

* Active Charcot arthropathy
* Unable to use NPWT at home
* Untreated bone or soft tissue infection
* Is pregnant or plans to become pregnant
* Is nursing or actively lactating
* Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including untreated schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years.
* Active alcohol or substance abuse in the opinion of the investigator that could impair the subject's ability to provide informed consent, participate in the study protocol or record study materials. Active alcohol (> 14 drinks per week over the last 3 months) or substance abuse (current use of cocaine, heroin, or methamphetamines or if drug or alcohol use will interfere with follow-up visits in foot clinic in the opinion of the investigator

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | 12 weeks
  The primary objective of this trial is to evaluate the incidence of wound closure. Closure is defined as complete epithelialization with no drainage.

SECONDARY OUTCOMES:
Time to wound healing | 12 weeks
  Days to complete closure. Closure is defined as complete epithelialization with no drainage.
Differences in wound healing trajectories | 12 weeks
  Defined as the change in wound area per week. Measured by wound measuring camera and PI observation/physical exam. Reported as mm^2 per day.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No